CLINICAL TRIAL: NCT00830349
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Risperidone 1 mg Tablets and Risperdal 1 mg Tablets Administered as a 1 x 1 mg Tablet in Healthy Subjects Under Fasting Conditions
Brief Title: Risperidone 1 mg Tablet in Healthy Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 01172
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Risperidone

ARMS (2):
- 1 (Experimental): Risperidone 1 mg Tablets
  Interventions: Drug: Risperidone
- 2 (Active Comparator): Risperdal® 1 mg Tablets
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — 1 mg Tablet
  Arms: 1
Drug: Risperidone — 1 mg Tablets
  Other Names: Risperdal®
  Arms: 2

SUMMARY:
The objective of this study was to compare the rate and extent of absorption of risperidone 1 mg tablets (test) versus Risperdal® (reference) administered as a 1 x 1 mg tablet under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria

* Subjects will be females and/or males, non-smokers, 18 years of age and older.
* Subjects should read, sign and date an Informed Consent Form prior to any study procedure.
* Female Subjects will be post-menopausal or surgically sterilezed.
* Post-menopausal status is defined as absence of menses for the past 12 months,
* Sterile status is defined as hysterectomy, bilateral oophorectomy or tubal ligation at least 6 months ago.

Exclusion Criteria

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any history or presence of significant Neurological, hepatic, renal, endocrine, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Subjects who do not tolerate venipuncture.
* Positive urine drug screen at screening.
* Subjects who use tobacco in any form will not be eligible to participate in this study. Three months abstinence before screening is required.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG abnormalities (clinically significant) (PR interval greater than 225 msec or QTc segment greater than 450 msec) or vital sign abnormalities (systolic blood pressure lower than 100 or over 160 mmHg, or diastolic blood pressure lower than 60 or over 96; or heart rate less than 60 bpm) at screening.
* Subjects with BMI ≥30.0.
* History of seizures or other predisposing factors.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day (1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana, pot) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
* History of cardiac disease or family history of cardiac disease.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical subinvestigator, contraindicates the subject's participation in this study.
* History of allergic reactions to risperidone.
* Use of any drugs known to induce or inhibit hepatic drug metabolism, use of an investigational drug or participation on an investigation study within 30 days prior to the administration of the study medication.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Donation of plasma (500 mL) within 7 days or donation or significant loss of whole blood (500 mL) within 56 days prior to administration of the study medication.
* Positive alcohol breath test at screening.

Additional exclusion criteria for female subjects only:

o Positive urine pregnancy test at screening (performed on all females).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2001-06; Primary Completion 2001-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, MD, Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada